CLINICAL TRIAL: NCT04178044
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalated Phase Ⅰ Study to Evaluate the Safety, Tolerability, Pharmacokinetic(PK) and Pharmacodynamic(PD) of GB223 in Healthy Adult Subjects.
Brief Title: Phase Ⅰ Clinical Study Protocol of GB223 Monoclonal Antibody Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB223-001; V2.3; 16 Jan 2019
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Bone Tumor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GB223-group 1 (Experimental): Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:7mg/kg,single dose administration; 2 subjects receive placebo.
  Interventions: Biological: GB223,7mg/kg
- GB223-group 2 (Experimental): 21mg/kg
  Interventions: Biological: GB223,21mg/kg
- GB223-group 3 (Experimental): 63mg/kg
  Interventions: Biological: GB223,63mg/kg
- GB223-group 4 (Experimental): 119mg/kg
  Interventions: Biological: GB223,119mg/kg
- GB223-group 5 (Experimental): 140mg/kg
  Interventions: Biological: GB223,140mg/kg

INTERVENTIONS:
Biological: GB223,7mg/kg — Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:7mg/kg 2 subjects receive placebo.
  Other Names: Placebo
  Arms: GB223-group 1
Biological: GB223,21mg/kg — Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:21mg/kg 2 subjects receive placebo. The next dose group can be initiated only after the safety and tolerability are confirmed within 4 or 8 weeks after the previous dose is given.
  Other Names: Placebo
  Arms: GB223-group 2
Biological: GB223,63mg/kg — Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:63mg/kg 2 subjects receive placebo. The next dose group can be initiated only after the safety and tolerability are confirmed within 4 or 8 weeks after the previous dose is given.
  Other Names: Placebo
  Arms: GB223-group 3
Biological: GB223,119mg/kg — Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:119mg/kg 2 subjects receive placebo. The next dose group can be initiated only after the safety and tolerability are confirmed within 4 or 8 weeks after the previous dose is given.
  Other Names: Placebo
  Arms: GB223-group 4
Biological: GB223,140mg/kg — Injection; strength of 70mg/1ml/vial; subcutaneous injection; GB223:140mg/kg 2 subjects receive placebo. The next dose group can be initiated only after the safety and tolerability are confirmed within 4 or 8 weeks after the previous dose is given.
  Other Names: Placebo
  Arms: GB223-group 5

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability and pharmacokinetic (PK) profiles of single dose of GB223 in healthy subjects; the secondary objective is to evaluate the immunogenicity and pharmacodynamic (PD) profiles of single dose of GB223 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and contents, and voluntarily sign the informed consent form;
2. Aged from 18 to 65 years at ICF signing (inclusive), males or females;
3. At screening, the male body weight≥50kg, female body weight ≥45kg, the body weight of males and females is not more than 75kg (inclusive), body mass index (BMI) is within the range between 19 and 24.0 (both inclusive);
4. The following tests are normal, or the abnormalities are not clinically significant at screening: physical examination, vital sign, laboratory tests, ECG test, chest radiography and CT tests of upper and middle abdomen, PPD test and CT test of oral cavity;
5. The subjects and their partners agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 12 months after the administration of investigational products.
6. The subjects can receive follow-up visits as scheduled, well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

1. Lactating and pregnant women;
2. Subjects who have pregnancy plan within 12 months;
3. Subjects who currently or previously have osteomyelitis or osteonecrosis of jaws, or subjects who plan to receive invasive dental surgery or jaw surgery, or subjects whose wounds are not cured after dental or oral surgeries;
4. Subjects who have clear medical history of central nervous system, cardiovascular, renal, hepatic, gastrointestinal, respiratory, metabolic system or subjects with other significant diseases; subjects who have medical history of psychiatric disorders; subjects with medical history of hypertension or screening systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg, which are clinically significant at the discretion of the investigators; subjects who have medical history of orthostatic hypotension;
5. Any of the following is met: allergic constitution; known allergic to the components of the investigational product or allergy history to any drug or food or pollen; subjects who have abnormal serum immunoglobulin E (IgE) test;
6. Any of the current symptoms, signs or laboratory test abnormalities indicating the possible presence of acute or subacute infection (e.g., pyrexia, cough, urgent micturition, urodynia, abdominal pain, diarrhea, cutaneous infected wound etc.)
7. Subjects who have medical history of drug addiction or drug abuse;
8. Smoking more than 5 cigarettes/day or equivalent tobacco; or subjects who cannot stop smoking during the study period;
9. Weekly alcohol consumption more than 28 units (1 unit = 285 mL of beer or 25 mL of spirits or 100 mL of wine); or subjects who have positive breath alcohol test within 24 hours before the use of investigational drug;
10. Subjects who meet any of the following criteria: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5xULN, serum creatinine (Cr) > 1.0xULN;
11. Abnormal routine blood tests: any of the following is met: white blood cells (WBC)<3.0×109/L or >9.15×109/L, neutrophil count (ANC)<1.5×109/L, platelet count (PLT)<100×109/L, hemoglobin (HGB)<113g/L;
12. Abnormal serum calcium: current hypocalcaemia or hypercalcemia, or albumin-corrected serum calcium level is not within the normal laboratory range.
13. Any of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
14. Subjects with abnormal thyroid and parathyroid function and diseases affecting bone metabolism such as rheumatoid arthritis and osteomalacia;
15. Subjects with recent fracture (within 6 months);
16. Subjects with positive tumor markers (CEA, AFP, PSA and CA-125);
17. Patients who previously or currently have malignant tumors within 5 years before screening (excluding adequately treated and completely cured skin basal cell carcinoma or squamous cell carcinoma, cervical in situ carcinoma);
18. Participated in other clinical studies within 3 months before enrollment, or subjects who received drugs which are known to injure the major organs within 3 months before enrollment;
19. Participated in clinical studies of similar investigational products such as denosumab etc.;
20. Use of drugs which may affect bone metabolism within 4 weeks or 5 half-lives (whichever is longer) before this study and the use of drugs which may affect bone metabolism during this study period; These drugs include but are not limited to the following drugs: contraceptives containing estrogen, bisphosphonate, fluoride, hormone replacement therapies (i.e., tibolone, estrogen, estrogenic compounds such as raloxifen), calcitonin, strontium, parathyroid hormone or its derivatives, vitamin D supplements (>1000IU/day), glucocorticoids (use of inhaled or local glucocorticoid 2 weeks before enrollment), anabolic hormone drugs (e.g., metandienone, nandrolone phenylpropionate, hydroxymetholone, stanozolol, nandrolone decanoate, danazolum), calcitriol and diuretics;
21. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Effect, AE | Up to 252 days
  Adverse Effect, AE
Serious Adverse Effect, SAE | Up to 252 days
  Serious Adverse Effect, SAE
AUC0-t | Up to 252 days
  AUC0-t
Cmax | Up to 252 days
  Cmax
AUC0-∞ | Up to 252 days
  AUC0-∞
Tmax | Up to 252 days
  Tmax
Vz/F | Up to 252 days
  Vz/F
Ke | Up to 252 days
  Ke
MRT | Up to 252 days
  MRT
t1/2z | Up to 252 days
  t1/2z
CLz/F | Up to 252 days
  CLz/F

SECONDARY OUTCOMES:
AntiDrug Antibody, ADA | Up to 252 days
  AntiDrug Antibody, ADA

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Liu, Bachelor, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li C, Liu H, Liao Y, Zhu Y, Tian J, Wang X, Hu Z, Zhan Y, Li X, Liang X, He J, Li Y, Shang D, Zheng Q, Wang T, Song H, Fang Y. Phase I, Randomized, Placebo-Controlled, Dose-Escalation Study of GB223, a Fully-Humanized Monoclonal Antibody to RANKL, in Healthy Chinese Adults. BioDrugs. 2023 Sep;37(5):721-735. doi: 10.1007/s40259-023-00604-7. Epub 2023 Jun 6. PMID 37278972